CLINICAL TRIAL: NCT00221052
Title: Relation Between Reduction of the Inflammatory Status and Glucose Metabolism in Healthy Overweight Men
Brief Title: Effect of Reduction of Inflammatory Status on Glucose Metabolism in Overweight Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: TNO-P6374
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-10

CONDITIONS: Overweight; Obesity; Inflammation
MeSH Terms: conditions — Overweight; Obesity; Inflammation | interventions — Diclofenac

INTERVENTIONS:
Drug: Diclofenac

SUMMARY:
Overweight increases the risk to develop chronic diseases including type-2 diabetes and cardiovascular disease. The low-grade inflammatory status often seen in overweight subjects is thought to play an important role in disease development.

The purpose of this study is to determine the role of inflammation on glucose metabolism and insulin resistance. In this study the effect of the anti-inflammatory treatment diclofenac on markers of inflammation and on parameters of glucose metabolism will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI): 25.1 - 32.0 kg/m2
* Normal Dutch eating habits

Exclusion Criteria:

* diabetes, cardiovascular disease or hypertension
* Not suitable to receive diclofenac treatment
* Smoking
* Extreme physical activity (more than 6 hours/week)
* Reported slimming or medically prescribed diet

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-06; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Trinette van Vliet, PhD, Principal Investigator — TNO Quality of Life, Location Zeist
Locations (1):
- TNO Quality of Life, Zeist, Netherlands

REFERENCES:
- [Derived] van Erk MJ, Wopereis S, Rubingh C, van Vliet T, Verheij E, Cnubben NH, Pedersen TL, Newman JW, Smilde AK, van der Greef J, Hendriks HF, van Ommen B. Insight in modulation of inflammation in response to diclofenac intervention: a human intervention study. BMC Med Genomics. 2010 Feb 23;3:5. doi: 10.1186/1755-8794-3-5. PMID 20178593